CLINICAL TRIAL: NCT07013526
Title: Dexmedetomidine as Adjuvant for Suprazygomatic Maxillary Nerve Block in Children's Adenotonsillectomy: a Randomized Controlled Trial Study
Brief Title: Dexmedetomidine as Adjuvant for Suprazygomatic Maxillary Nerve Block in Children's Adenotonsillectomy
Acronym: SZMB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Gianluca Bertolizio, Dr, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2026-11731
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Adenotonsillectomy
Keywords: pain; opioid-free recovery; Suprazygomatic maxillary nerve block
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group R (Other): Group R will receive an SZMB of 0.15 ml/kg of local anesthetic ropivacaine 0.2% (max 5 ml). After the block, 0.1 ml/kg of normal saline will be administered intravenously. No dexmedetomidine will be given.
  Interventions: Procedure: Ropivacaine
- Group RD (Experimental): 2. Group RD will receive an SZMB of 0.1 ml/kg of a solution of local anesthetic ropivacaine 0.2% and dexmedetomidine 1 mcg/ml (max 5 ml). After the block, 0.1 ml/kg of normal saline will be administered intravenously. No dexmedetomidine i.v. will be given.
  Interventions: Procedure: Ropivacaine
- Group D (Other): Group D will receive an SMB of 0.1 ml/kg of local anesthetic ropivacaine 0.2% (max 5 ml). After the block a bolus of intravenous dexmedetomidine 0.25 mcg/kg i.v. will be given.
  Interventions: Procedure: Ropivacaine

INTERVENTIONS:
Procedure: Ropivacaine — Administration of ropivacaine in a Suprazygomatic maxillary nerve block

SUMMARY:
The goal of this clinic trial is to evaluate the impact of dexmedetomidine as an adjunct pain pain medication on opioid-free recovery in children undergoing adenotonsillectomy with Suprazygomatic maxillary nerve block (SZMB). The main questions it aims to answer are:

* Does SZMB with the local anesthetic ropivacaine and the adjuvant dexmedetomidine result in less pain
* Is dexmedetomidine associated with an improved quality of recovery at home Researchers will compare pain in participants given an SZMB with ropivacaine and an adjuvant dexmedetomidine, participants given SZMB with ropivacaine only, and a SZMB with ropivacaine and dexmedetomidine given intravenously.

Participants will:

* Be given the SZMB during the surgery.
* Be evaluated after surgery to measure their opioid consumption, pain severity, level of agitation, and level of delirium
* Complete a daily questionnaire for 7 days after surgery on the patients pain and recovery

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective partial adenotonsillectomy,
* STUBR score ≥ 3, indicating significant sleep-disordered breathing
* Patients whose parents are fluent in French of English will be enrolled

Exclusion Criteria:

* Scheduled to undergo total extracapsular adenotonsillectomy or adenoidectomy-only procedures
* Patient requires prolonged intubation postoperatively
* the anesthesiologist does not adhere to the standardized anesthesia protocol
* Patients with neurological or cardiac congenital deficits, with cardiac arrhythmias (non-sinus rhythm), implanted pacemakers, on chronic therapy with drugs that have known effects on sympathetic and parasympathetic activity (antimuscarinics, beta-2 adrenergic agonists, alpha-1 adrenergic antagonists or antiarrhythmic agents, tricyclic antidepressants)
* ASA physical status III or higher
* Parent/legal guardians refuses to participate
* Patients scheduled for surgery without an appointment at the Montreal Children's Hospital (MCH) Preoperative Clinic will not be enrolled in the study.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Opioid-free recovery | 2 hours
  Incidence of patients not requiring opioids in the PACU after surgery

SECONDARY OUTCOMES:
Number of patients with postoperative Pain | 2 hours
  Patients were classified as having pain if they had a Face, Activity, Cry, Consolability (FLACC) score that was greater than or equal to 3.
Number of Patients with Emergence Delirium | 2 hours
  Patients were classified as having emergence delirium if they had a score on the emergence delirium scale that was greater than or equal to 10 in the Post-anesthesia care unit.
Pain through follow-up | 7 days
  Difference in pain between the groups, assessed with the Parents' Postoperative Pain Measure
Quality of Recovery through follow-up | 7 days
  Differences in the Quality of recovery between the groups, as measured by the Post-Hospitalization Behavior Questionnaire for Ambulatory Surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No